CLINICAL TRIAL: NCT04122937
Title: Molecular Characterisation and Clinical Implications of Inflammation Related to Peritoneal Carcinomatosis in Women With Ovarian or Colon Cancer.
Brief Title: Defining Inflammation Related to Peritoneal Carcinomatosis in Women With Ovarian or Colon Cancer.
Acronym: CarFlog
Status: Completed | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Anna Solini, Associate Professor, University of Pisa
Other Study IDs: AS0003
Record Dates: First submitted 2019-10-09; First posted 2019-10-10 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Peritoneal Carcinomatosis; Ovarian Cancer; Colon Cancer
Keywords: peritoneal carcinomatosis; colon cancer; ovarian cancer; P2X7R-inflammasome
MeSH Terms: conditions — Peritoneal Neoplasms; Ovarian Neoplasms; Colonic Neoplasms | interventions — Cytoreduction Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — peritoneal biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ovarian cancer: Patients affected by ovarian cancer will be stratified according to BRCA1 and BRCA2 mutational status.
  Interventions: Procedure: Cytoreductive surgery
- Colon cancer: Patients affected by colon cancer will be similarly stratified according to BRAF and KRAS mutational status and to the presence of low-grade or high-grade microsatellite instability (MSI).
  Interventions: Procedure: Cytoreductive surgery

INTERVENTIONS:
Procedure: Cytoreductive surgery — Partial removal of peritoneal tissue involved by neoplastic invasion
  Other Names: Debulking

SUMMARY:
Inflammation plays an important role in the pathogenesis of peritoneal carcinosis. Patients with elevated levels of different inflammation cytokines show a worse prognosis at the time of diagnosis. In women, ovarian and colon cancer are the main causes of peritoneal carcinosis and a comparison of these two different types of peritoneal invasion have not been conducted yet. We found interesting studying the role of immune response, in particular tumour-associated antigens (TAA) that modulate the metastatic process. We will investigate also mitochondrial defects, such as mutations in mt-DNA, potentially involved in carcinogenesis.

DETAILED DESCRIPTION:
At the time of hospitalization all the patients will undergo a complete clinical evaluation with determination of biochemical parameters such as fasting blood glucose, blood count, hs-CRP, AST and ALT, uric acid, creatinine and BUN. An extra blood aliquot will be collected to assess the serum biomarkers under investigation.

During surgery two samples of peritoneal tissue macroscopically undamaged will be collected. On those samples will be executed separation of adipocytes cells, RNA and protein extraction for measuring of inflammatory and neoplastic biomarkers, determination of P2X7R-inflammasome activity and mitochondrial DNA analyse.

ELIGIBILITY:
Inclusion Criteria:

* histological diagnosis of peritoneal carcinosis secondary to colon cancer or high-grade ovarian cancer
* patients able to consent

Exclusion Criteria:

* previous malignancies, except for patients with cutaneous basal cell carcinoma, Cervical Intraepithelial Neoplasia (CIN) or melanoma in situ
* current chemotherapy or radiotherapy
* current steroid therapy or immunotherapy
* patients affected by systemic inflammatory disease and/or Inflammatory bowel disease (IBD)

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study consecutively enrolled 30 patients undergoing surgical treatment for peritoneal carcinosis: 15 patients affected by high grade ovarian cancer and 15 patients affected by colon cancer. Patients will be enrolled among those referring to the Gynaecologic Unit and the General Surgery Unit, University Hospital of Pisa, Italy.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Immune biomarkers level | Each patients will be assessed at baseline
  Serum level of different immune related biomarkers (such as CD4, CD8, CUZD1, LAG3, PD1, PDL1, IMP1 and p62/IMP2) will be determined using ELISA.
Metastatic mediators level | Each patients will be assessed at baseline
  Peritoneal expression of cytokines related to metastatic process (such as IL6, IL2, TNFα, TGFβ1, VEGF, CD68, FGFR1, CCL2/MCP-1, CD73) will be determined using real time-PCR.
P2X7R-inflammasome activity | Each patients will be assessed at baseline
  Peritoneal expression of NLRP3-ASC will be determine using RT-PCR

CONTACTS AND LOCATIONS:
Overall Officials: Anna Solini, MD, PhD, Principal Investigator — University of Pisa
Locations (1):
- University of Pisa, Pisa, Italy